CLINICAL TRIAL: NCT03552744
Title: Colorectal Cancer Testing in Swiss Primary Care: A Cluster Randomized Controlled Trial Among Primary Care Physicians of the Swiss Sentinel Surveillance Network
Brief Title: Colorectal Cancer Screening Among Primary Care Physicians of the Swiss Sentinel Surveillance Network
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: RCTSentinella2018
Record Dates: First submitted 2018-05-25; First posted 2018-06-12 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: Mailed training intervention
- Control group (No Intervention)

INTERVENTIONS:
Other: Mailed training intervention — PCPs from the intervention group will be mailed an intervention package that includes:
  1. 2-page structured evidence summary on CRC screening and information about Colonoscopy & FIT ("Decision box")
  2. patient decision aid (20-page booklet) on CRC screening for distribution to patients (Decision Aid)
  3. video example for the PCP, which illustrates a participatory approach to discussing CRC screening with a patient
  4. 4-page abridged version of the booklet to support PCPs when they discuss CRC screening with patients during a clinical visit ("Decision Board")
  5. individualized 1-page summary of PCP screening practices comparing their individual prescription patterns to group patterns, based on the data collected in 2017 ("Performance card")
  6. 2-page document that encourages PCPs still using the inferior guaiac-based FOBT to switch to FIT and includes list of laboratories from which they can order FIT
  7. sample FIT for PCPs who may not be familiar with its contents and use
  Arms: Intervention group

SUMMARY:
Colorectal cancer (CRC) is the third leading cause of cancer mortality in Switzerland, and kills 1600 people annually. Most deaths could be prevented by screening, but the 2012 Swiss national health survey found that only 40% of 50-75-year-olds had been tested within recommended intervals (26% with colonoscopy in the last 10 year, 7% with fecal occult blood test [FOBT] in the last 2 years, and 7% with both). If screening starts at age 50, in the average risk population absolute risk of dying from CRC at age 80 can be cut from 2% to 1%, reducing relative risk by 50%. Since 2013, Switzerland has reimbursed screening by colonoscopy every 10 years or FOBT every 2 years for adults 50-69 years old. Conforming to current recommendations, the Federal Office of Public Health (FOPH) officially recognizes both screening modalities.

When patients are offered a choice of screening test (colonoscopy vs. FOBT), they are as likely to opt for one as the other. Patient preferences are unlikely to vary much between PCP practices, so distribution of colonoscopy and FOBT within each practice should also be roughly equal. Family physicians are recognized as the most trusted professional to discuss CRC screening in Switzerland. However, many primary care physicians (PCPs) prefer prescribing colonoscopy over FOBT, but physician preference for method seems to vary widely between regions. If physician preferences and local medical culture currently influence choice of method more strongly than patient preferences, encouraging PCPs to diagnose patient preferences for screening method may reduce the number of PCPs who prescribe only one method. An earlier study in Switzerland showed that training PCPs and giving them educational support and decision aids raised the number who intend to prescribe colonoscopy and FOBT in equal proportions. A randomized controlled trial in the US showed that when patients were offered both FOBT and colonoscopy rather than only colonoscopy alone, more patients were screened for CRC. Offering choice of method may thus increase overall screening rates.

The Swiss Sentinel Surveillance Network (Sentinella) is a cooperative surveillance project including the Federal Office of Public Health (FOPH), PCPs representatives and the five Swiss institutes of family medicine. A sample of 150 to 250 general practitioners, internists and pediatricians in private practices from all regions of Switzerland report weekly morbidity data to the network using irreversibly anonymized patient data collected during consultations. In 2017, 91 out of 129 eligible PCPs of the Sentinella network participated in a cross-sectional data collection on CRC screening. The Sentinella network appears ideally suited to perform an intervention in order to modify screening practices and measure outcomes using the same collection form as in 2017.

This study will test the benefits of a prepackaged training program in participatory medicine sent by post to PCPs in Switzerland. The package is designed to improve their diagnoses of patient preferences for screening and screening method (colonoscopy or FOBT). The study begins with the hypothesis that giving PCPs evidence summaries on CRC screening, decision aids for patients, and performance feedback on the 2017 data collection will increase the number of PCPs whose patients include at least one screened with FOBT, and who will prescribe at least one FOBT/FIT (Fecal Immunochemical Test) instead of prescribing only colonoscopy. This might reduce variation in care between PCP practices by increasing variation in methods of screening prescribed within each PCP practices. Analyses from the 2017 data collection suggest that fewer patients refused CRC testing in practices that offered both methods than in practices that offered only colonoscopy. This intervention might increase screening rates overall, while respecting patient's autonomy to refuse the test and to be prescribed the test they prefer.

The study will compare outcomes among PCPs allocated to the intervention group to those in the control group, and will be measured by collecting anonymous structured patient data on 40 consecutive patients by PCPs and questionnaires filled by PCPs.

The study is designed to fit within the Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM) framework for structuring data collection. RE-AIM ensures that a study's outcomes for future implementation and dissemination works are collected. The RE-AIM criteria will be used to identify the translatability and public health impact of this intervention, and for making clear to future stakeholders the internal and external validity of study results.

ELIGIBILITY:
Inclusion Criteria:

* Physician-level: PCPs participating in the Swiss Sentinel Surveillance Network (Sentinella) willing to participate in the study
* Patient-level: Each PCP will collect data on 40 consecutive patients aged 50 to 75 years old seen in PCP offices over a 2 weeks to 2 months period. Patients will be included if there is a face-to-face consultation billed for at least 5 minutes at the practice.

Exclusion Criteria:

* None except criteria which do not respect inclusion criteria

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Number of PCPs who have at least one patient ever tested with FOBT, or who prescribe at least one FOBT to eligible patients (patients not already tested within recommended intervals, with no contra-indication for screening). | At 3 months after intervention
  PCPs systematically collect data from 40 consecutive patients, aged 50-75 years

SECONDARY OUTCOMES:
Number of PCPs whose proportion of patients previously tested or planning to be tested with FOBT/colonoscopy is at least 40% (the PCP must have discussed screening with these patients, who have no symptoms or risk factors for CRC | At 3 months after intervention
  PCPs systematically collect data from 40 consecutive patients, aged 50-75 years
Number of PCPs who discussed CRC with >50% of their eligible patients (patients not tested within recommended intervals, with no contra-indications for CRC screening) | At 3 months after intervention
  PCPs systematically collect data from 40 consecutive patients, aged 50-75 years
Change in PCPs' future intentions to prescribe CRC screening tests | At 3 months after intervention
  A questionnaire completed by participating PCPs
Change in PCPs' future intentions to prescribe colonoscopy vs. FOBT over the next 6 months | At 3 months after intervention
  A questionnaire completed by participating PCPs

CONTACTS AND LOCATIONS:
Overall Officials: Reto Auer, MD, MAS, Principal Investigator — Institute of primary health care (BIHAM), University of Bern
Locations (1):
- Institute of Primary Health Care (BIHAM), University of Bern, Bern, Switzerland

REFERENCES:
- [Background] Meester RG, Doubeni CA, Lansdorp-Vogelaar I, Goede SL, Levin TR, Quinn VP, Ballegooijen Mv, Corley DA, Zauber AG. Colorectal cancer deaths attributable to nonuse of screening in the United States. Ann Epidemiol. 2015 Mar;25(3):208-213.e1. doi: 10.1016/j.annepidem.2014.11.011. Epub 2014 Dec 5. PMID 25721748
- [Background] Fedewa SA, Cullati S, Bouchardy C, Welle I, Burton-Jeangros C, Manor O, Courvoisier DS, Guessous I. Colorectal Cancer Screening in Switzerland: Cross-Sectional Trends (2007-2012) in Socioeconomic Disparities. PLoS One. 2015 Jul 6;10(7):e0131205. doi: 10.1371/journal.pone.0131205. eCollection 2015. PMID 26147803
- [Background] Gigerenzer G. Towards a paradigm shift in cancer screening: informed citizens instead of greater participation. BMJ. 2015 May 5;350:h2175. doi: 10.1136/bmj.h2175. No abstract available. PMID 25943239
- [Background] Schroy PC 3rd, Emmons KM, Peters E, Glick JT, Robinson PA, Lydotes MA, Mylvaganam SR, Coe AM, Chen CA, Chaisson CE, Pignone MP, Prout MN, Davidson PK, Heeren TC. Aid-assisted decision making and colorectal cancer screening: a randomized controlled trial. Am J Prev Med. 2012 Dec;43(6):573-83. doi: 10.1016/j.amepre.2012.08.018. PMID 23159252
- [Background] European guidelines for quality assurance in colorectal cancer screening and diagnosis. Luxembourg: Publications Office of the European Union, 2012
- [Background] publique, O.f.d.l.s., Dépistage du cancer du côlon. 2013: p. p. 455
- [Background] Bulliard JL, Ducros C, Levi F. [Organized screening for colorectal cancer: challenges and issues for a Swiss pilot study]. Rev Med Suisse. 2012 Jul 11;8(348):1464-7. French. PMID 22934475
- [Background] Klabunde CN, Lanier D, Nadel MR, McLeod C, Yuan G, Vernon SW. Colorectal cancer screening by primary care physicians: recommendations and practices, 2006-2007. Am J Prev Med. 2009 Jul;37(1):8-16. doi: 10.1016/j.amepre.2009.03.008. Epub 2009 May 13. PMID 19442479
- [Background] McQueen A, Bartholomew LK, Greisinger AJ, Medina GG, Hawley ST, Haidet P, Bettencourt JL, Shokar NK, Ling BS, Vernon SW. Behind closed doors: physician-patient discussions about colorectal cancer screening. J Gen Intern Med. 2009 Nov;24(11):1228-35. doi: 10.1007/s11606-009-1108-4. Epub 2009 Sep 18. PMID 19763699
- [Background] Meissner HI, Breen N, Klabunde CN, Vernon SW. Patterns of colorectal cancer screening uptake among men and women in the United States. Cancer Epidemiol Biomarkers Prev. 2006 Feb;15(2):389-94. doi: 10.1158/1055-9965.EPI-05-0678. PMID 16492934
- [Background] Cooper GS, Koroukian SM. Geographic variation among Medicare beneficiaries in the use of colorectal carcinoma screening procedures. Am J Gastroenterol. 2004 Aug;99(8):1544-50. doi: 10.1111/j.1572-0241.2004.30902.x. PMID 15307875
- [Background] Wennberg JE. Unwarranted variations in healthcare delivery: implications for academic medical centres. BMJ. 2002 Oct 26;325(7370):961-4. doi: 10.1136/bmj.325.7370.961. No abstract available. PMID 12399352
- [Background] Mulley AG, Trimble C, Elwyn G. Stop the silent misdiagnosis: patients' preferences matter. BMJ. 2012 Nov 8;345:e6572. doi: 10.1136/bmj.e6572. No abstract available. PMID 23137819
- [Background] Selby K, Cornuz J, Gachoud D, Bulliard JL, Nichita C, Dorta G, Ducros C, Auer R. Training primary care physicians to offer their patients faecal occult blood testing and colonoscopy for colorectal cancer screening on an equal basis: a pilot intervention with before-after and parallel group surveys. BMJ Open. 2016 May 13;6(5):e011086. doi: 10.1136/bmjopen-2016-011086. PMID 27178977
- [Background] Inadomi JM, Vijan S, Janz NK, Fagerlin A, Thomas JP, Lin YV, Munoz R, Lau C, Somsouk M, El-Nachef N, Hayward RA. Adherence to colorectal cancer screening: a randomized clinical trial of competing strategies. Arch Intern Med. 2012 Apr 9;172(7):575-82. doi: 10.1001/archinternmed.2012.332. PMID 22493463
- [Background] Hurlimann D, Limacher A, Schabel M, Zanetti G, Berger C, Muhlemann K, Kronenberg A; Swiss Sentinel Working Group. Improvement of antibiotic prescription in outpatient care: a cluster-randomized intervention study using a sentinel surveillance network of physicians. J Antimicrob Chemother. 2015 Feb;70(2):602-8. doi: 10.1093/jac/dku394. Epub 2014 Oct 17. PMID 25326088
- [Background] Glasgow RE. RE-AIMing research for application: ways to improve evidence for family medicine. J Am Board Fam Med. 2006 Jan-Feb;19(1):11-9. doi: 10.3122/jabfm.19.1.11. PMID 16492000